CLINICAL TRIAL: NCT05994508
Title: A Community Pickleball Program for People With Parkinson Disease: A Feasibility and Preliminary Results Study
Brief Title: Feasibility and Effects of a Pickleball Program for People With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwestern University (Other)
Collaborators: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRBAZ/5214
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): A single group of participants with Parkinson disease will participate in a 6-week pickleball program with pre-test, post-test, and one month follow-up testing.
  Interventions: Other: Pickleball program

INTERVENTIONS:
Other: Pickleball program — The intervention will be a 6-week pickleball program, at a frequency of two times a week. Each session will be one hour which will consist of dynamic warm-up drills, pickleball-related skill practice and game play, and a cool-down period.

SUMMARY:
Pickleball is a fast-growing sport that has been shown to improve social integration, life satisfaction, function, and cognitive function in older adults. Parkinson disease is a neurodegenerative disorder characterized by bradykinesia, rigidity, tremors, and postural instability. Exercise has been shown to improve physical and cognitive function in people with Parkinson disease (PD). The purpose of this study is to assess if a community pickleball program can be a feasible and effective for people living with PD.The primary aim of this study is to assess the feasibility of a group pickleball program for people with PD. Secondary aims is to assess the effects of a 6-week pickleball exercise program on balance, gait, cognition, upper extremity function, pain, and quality of life in people with PD. This will be a pre-test, post-test single-group, prospective, mixed-methods study with 1- month follow-up. Sixteen participants will be enrolled in a 6-week pickleball program, at a frequency of twice a week for one hour each session. Feasibility will be assessed by retention rates, adherence rates, resources, and number of adverse events. Quantitative data to be collected will include the Mini-BESTest, gait and body posture variables, Parkinson's Disease Questionnaire-8, the Shirt-Buttoning Task, 9 Hole Peg Test, grip strength, PD-Pain Classification System, and the National Institutes of Health Toolbox Cognition Battery. Additionally, participants will be scheduled for small semi-structured focus group interviews to gain qualitative data about their experiences of the program. It is hypothesized that a pickleball program for people living with PD will be a feasible activity and will result in improvements in balance, gait, cognition, upper extremity function, and quality of life. Additionally, it is hypothesized that participants will have a favorable opinion on the activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson disease
* Able to walk without an assistive device
* Able to tolerate 45 minutes of activity with occasional seated rest

Exclusion Criteria:

* Diagnosis of any other neurologic disorder
* Any current illness, injury, or cognitive function that would prevent ability to perform the study tasks
* Not regularly participating in pickleball (less than 3 times a month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Mini-BEStest | Within 7 day before and after the intervention as well as one-month after intervention completion
  Comprehensive balance assessment
10-Meter Walk Test | Within 7 day before and after the intervention as well as one-month after intervention completion
  Measure of gait speed
Grip strength dynamometry | Within 7 day before and after the intervention as well as one-month after intervention completion
  Assessment of grip strength

SECONDARY OUTCOMES:
The shirt-buttoning task | Within 7 day before and after the intervention as well as one-month after intervention completion
  An upper limb functional performance test
9-Hole Peg Test | Within 7 day before and after the intervention as well as one-month after intervention completion
  Assessment of finger dexterity
Parkinson's Disease Questionnaire-8 | Within 7 day before and after the intervention as well as one-month after intervention completion
  Measure of perceived quality of life. Scores range from 0% to 100% with higher scores representing greater impact of the disease.
Montreal Cognitive Assessment | Within 7 day before and after the intervention as well as one-month after intervention completion
  Assessment of cognitive abilities scored on a scale from 0-30. Higher scores represent higher cognitive abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne O'Neal, DPT, DHSc, Principal Investigator — Midwestern University
Locations (1):
- Creighton University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No